CLINICAL TRIAL: NCT06033807
Title: Active Screening of Latent Tuberculosis Infection in School Contacts of Active Tuberculosis Patients
Status: Recruiting | Type: Observational
Sponsor: Huashan Hospital (Other)
Collaborators: Guizhou Center for Disease Control and Prevention (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Professor, Huashan Hospital
Other Study IDs: TB-Youth Screening
Record Dates: First submitted 2023-08-29; First posted 2023-09-13 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Tuberculosis; Latent Tuberculosis Infection
Keywords: latent tuberculosis; active screening
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Contacts: School contacts of ATB patients
  Interventions: Diagnostic Test: QuantiFERON-TB Gold (QFT) test

INTERVENTIONS:
Diagnostic Test: QuantiFERON-TB Gold (QFT) test — Participants will be tested by QuantiFERON-TB Gold (QFT) test to see if they have ever infected by MTB. Those with positive results will proceed to sputum Xpert MTB/RIF, physical examination and chest CT scan, as well as sputum culture if necessary to distinguish latent TB infection (LTBI) from ATB. X-ray scan is conditional on age above 15 years with a positive QuantiFERON-TB Gold (QFT) test result.
  Other Names: Chest CT Scan; Chest X-ray Scan; Sputum Culture; Sputum Xpert MTB/RIF

SUMMARY:
The goal of this observational study is to investigate the proportion of Mycobacterium tuberculosis (MTB) infection in school contacts of active tuberculosis (ATB) patients. The main questions it aims to answer are:

* the proportion of MTB infection among school contacts of ATB patients
* risk factors related to tuberculosis (TB) infection
* health economic evaluation of screening strategy

ELIGIBILITY:
Inclusion Criteria:

* 13 years old or above;
* Students in junior middle school, high school and university;
* Close contact of school active tuberculosis case (e.g. in the same classroom, in the same dormitory);
* Himself/herself (together with his/her guardian for age under 18 years old) willing to participate in trial and sign informed consent.

Exclusion Criteria:

* Current clinical or sputum culture confirmed active tuberculosis
* Have completed a full course of treatment for ATB or LTBI

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Students in junior middle schools, high schools and universities from Guizhou Province, China
Sampling Method: Probability Sample
Enrollment: 31440 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of tuberculosis (TB) infection in school contacts | baseline
  The prevalence of TB infection is defined as the number of participants with positive results in QuantiFERON-TB Gold (QFT) test in study population. Positive result in QFT test indicates higher response than the cut-off value of 0.35 IU / ml of INF-γ detected in at least one test tube (TB1 or TB2).

SECONDARY OUTCOMES:
Age | baseline
  Age as possible risk factor of tuberculosis infection
Sex | baseline
  Sex as possible risk factor of tuberculosis infection.
Vaccination history checklist | baseline
  Bacillus Calmette-Guérin (BCG) vaccination history as possible risk factor of tuberculosis infection.
Patterns of contacting checklist | baseline
  Duration, size of space of exposure to active tuberculosis-infected patient; as possible risk factor of tuberculosis infection.
Co-morbidities / medical history checklist | baseline
  Co-morbidities / medical history [cardiovascular disease, bronchial asthma, digestive ulcer, nephritic syndrome, glomerulonephritis, diabetes, hyperthyroidism, systemic lupus erythematosus, ankylosing spondylitis, epilepsy, schizophrenia, depression, HIV infection, glucocorticoid use, biologic agent use, immunosuppressive agent use, or other relevant co-morbidities / medical history]; as possible risk factor of tuberculosis infection.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, PhD, Principal Investigator — Huashan Hospital
Locations (44):
- China (44):
  - Xinpu New Area Center of Disease Control, Zunyi, Guiyang
  - Dafang Center for Disease Control and Prevention, Bijie, Guizhou
  - Qixingguan Center for Disease Control and Prevention, Bijie, Guizhou
  - Nayong Center for Disease Control and Prevention, Bijie, Guizhou
  - Hezhang Center for Disease Control, Bijie, Guizhou
  - Jinsha Center for Disease Control, Bijie, Guizhou
  - Qianxi Center of Disease Control, Bijie, Guizhou
  - Weining Center of Disease Control, Bijie, Guizhou
  - Zhijin Center of Disease Control, Bijie, Guizhou
  - Liping Center for Disease Control and Prevention, Linping, Guizhou
  - Liuzhi Special District Center of Disease Control, Liupanshui, Guizhou
  - Panzhou Center of Disease Control, Liupanshui, Guizhou
  - Shuicheng District Center of Disease Control, Liupanshui, Guizhou
  - Cengong Center of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Congjiang Ceter of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Danzhai Center of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Huangping Center of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Jianhe Center of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Jinping Center of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Kaili Center of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Leishan Center of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Majiang Center of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Rongjiang Center of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Sansui Center of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Shibing Center of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Taijiang Center of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Tianzhu Center of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Zhenyuan Center of Disease Control, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - Qingzhen Center for Disease Control and Prevention, Qingzhen, Guizhou
  - Bozhou District Center of Disease Control, Zunyi, Guizhou
  - Chishui Center of Disease Control, Zunyi, Guizhou
  - Daozhen Center of Disease Control, Zunyi, Guizhou
  - Fenggang Center of Disease Control, Zunyi, Guizhou
  - Honghuagang District Center of Disease Control, Zunyi, Guizhou
  - Huichuan District Center of Disease Control, Zunyi, Guizhou
  - Meitan Center of Disease Control, Zunyi, Guizhou
  - Renhuai Center of Disease Control, Zunyi, Guizhou
  - Suiyang Center of Disease Control, Zunyi, Guizhou
  - Tongzi Center of Disease Control, Zunyi, Guizhou
  - Wuchuan Center of Disease Control, Zunyi, Guizhou
  - Xishui Center of Disease Control, Zunyi, Guizhou
  - Yuqing Center of Disease Control, Zunyi, Guizhou
  - Zhengan Center of Disease Control, Zunyi, Guizhou
  - Dalian Public Health Clinical Center, Dalian, Liaoning

IPD SHARING:
Plan to Share IPD: No
This research targets adolescent students in school. We decide not to share IPD from the ethical perspective.